CLINICAL TRIAL: NCT00227747
Title: Randomized Phase III Trial Comparing in a Preoperative Schedule the Result of Two Concurrent Chemoradiation Schemes (45 Gy + Capecitabine vs 50 Gy + Capecitabine - Oxaliplatin) on the Rate of Sterilization of the Operative Specimen in Resectable Rectal Carcinomas T3-4 No-2 Mo
Brief Title: Radiation Therapy and Capecitabine With or Without Oxaliplatin in Treating Patients Who Are Undergoing Surgery for Stage II or Stage III Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445034; FRE-FNCLCC-ACCORD-12/0405; EU-20522
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Radiothérapie + Xelox (Experimental)
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy
- Radiothérapie + Capécitabine (Active Comparator)
  Interventions: Drug: capecitabine; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin
  Arms: Radiothérapie + Xelox
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving radiation therapy together with combination chemotherapy before surgery may shrink the tumor so it can be removed. It is not yet known whether giving radiation therapy together with capecitabine is more effective with or without oxaliplatin before surgery in treating rectal cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy, capecitabine, and oxaliplatin to see how well they work compared to radiation therapy and capecitabine in treating patients who are undergoing surgery for stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of neoadjuvant chemoradiotherapy comprising radiotherapy and capecitabine with vs without oxaliplatin followed by total mesorectal excision, in terms of the rate of complete surgical resection, in patients with resectable stage II or III rectal cancer.

Secondary

* Compare overall and disease-free survival of patients treated with these regimens.
* Compare clinical tumor response in patients treated with these regimens.
* Compare acute and late toxicity of these regimens in these patients.
* Determine biological parameters that predict tumor response and treatment-related toxicity in patients treated with these regimens.
* Compare sphincter preservation and function in patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily 5 days a week and receive capecitabine once daily 5 days a week in weeks 1-5.
* Arm II: Patient undergo radiotherapy and receive capecitabine as in arm I. Patients also receive oxaliplatin once weekly in weeks 1-5.

All patients undergo total mesorectal excision 6 weeks after completion of chemoradiotherapy.

PROJECTED ACCRUAL: A total of 590 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * T3-4, N0-2, M0 disease by endorectal ultrasound

    * T2 disease located in the low rectum allowed provided lower pole is ≤ 6 cm from the anal verge
* Tumor must be accessible to digital rectal examination (i.e., tumor located at low- or mid-rectum)
* Resectable disease treatable with chemoradiotherapy

  * No unresectable disease (i.e., T4 disease with high risk for incomplete gross resection [i.e., R2])

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* Alkaline phosphatase normal
* Bilirubin normal

Renal

* Creatinine ≤ 130 μmol/L
* No severe renal insufficiency

Cardiovascular

* No cardiac insufficiency
* No symptomatic coronary artery disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindication to study treatment
* Prior acute intestinal obstruction allowed provided patient underwent surgical diversion with stoma
* No history of other cancer except basal cell skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy
* No uncontrolled diabetes
* No other uncontrolled severe disease
* No geographical, social, or psychological condition that would preclude study follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for cancer
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for cancer

Surgery

* Not specified

Other

* No concurrent phenytoin
* No concurrent participation in another clinical trial of an experimental medical treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2005-11-08 (Actual); Primary Completion 2008-10-22 (Actual); Study Completion 2013-07-15 (Actual)

PRIMARY OUTCOMES:
Rate of complete surgical resection

SECONDARY OUTCOMES:
Overall survival
Disease-free survival
Sphincter preservation
Sphincter function
Biological parameters that predict tumor response and treatment-related toxicity
Acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Gerard, MD, Study Chair — Centre Antoine Lacassagne
Locations (69):
- France (69):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier, Altkirch
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Hopital de Beziers, Béziers
  - Centre Hospitalier de Blois, Blois
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Clinique Sainte Marie, Chalon-sur-Saône
  - Hopital Louis Pasteur, Chartres
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Drevon, Dijon
  - Hopital Du Bocage, Dijon
  - Centre Hospitalier de Gap, Gap
  - Clinique Sainte-Marguerite, Hyères
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Hopital Robert Boulin, Libourne
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Jean Bernard, Limoges
  - Centre Hospitalier General, Longjumeau
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Clinique J. B. Menis, Mâcon
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier General Andre Boulloche, Montbéliard
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Clinique Clementville, Montpellier
  - Clinique Plein Ciel, Mougins
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Clinique Hartmann, Neuilly-sur-Seine
  - Polyclinique du Val de Loire, Nevers
  - Centre Antoine Lacassagne, Nice
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier - Pau, Pau
  - Clinique Saint - Pierre, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - CHU - Robert Debre, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier de Rodez, Rodez
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Clinique Pasteur - Toulouse, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Centre d'Oncologie Saint-Yves, Vannes
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Gerard JP, Azria D, Gourgou-Bourgade S, Martel-Laffay I, Hennequin C, Etienne PL, Vendrely V, Francois E, de La Roche G, Bouche O, Mirabel X, Denis B, Mineur L, Berdah JF, Mahe MA, Becouarn Y, Dupuis O, Lledo G, Montoto-Grillot C, Conroy T. Comparison of two neoadjuvant chemoradiotherapy regimens for locally advanced rectal cancer: results of the phase III trial ACCORD 12/0405-Prodige 2. J Clin Oncol. 2010 Apr 1;28(10):1638-44. doi: 10.1200/JCO.2009.25.8376. Epub 2010 Mar 1. PMID 20194850
- [Derived] Azria D, Doyen J, Jarlier M, Martel-Lafay I, Hennequin C, Etienne P, Vendrely V, Francois E, de La Roche G, Bouche O, Mirabel X, Denis B, Mineur L, Berdah J, Mahe M, Becouarn Y, Dupuis O, Lledo G, Seitz J, Bedenne L, Gourgou-Bourgade S, Juzyna B, Conroy T, Gerard J. Late toxicities and clinical outcome at 5 years of the ACCORD 12/0405-PRODIGE 02 trial comparing two neoadjuvant chemoradiotherapy regimens for intermediate-risk rectal cancer. Ann Oncol. 2017 Oct 1;28(10):2436-2442. doi: 10.1093/annonc/mdx351. PMID 28961836